CLINICAL TRIAL: NCT04719546
Title: Identifying Risk Factors of Necrotizing Enterocolitis in the NICU of Nancy Benchmarking With the NICU of Lyon Over 10 Years
Brief Title: Risk Factors of Necrotizing Enterocolitis in Premature Newborns
Acronym: ECUNancyLyon
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Jean-Michel HASCOET, Professor, Central Hospital, Nancy, France
Other Study IDs: 2020PI279
Record Dates: First submitted 2021-01-14; First posted 2021-01-22 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Necrotizing Enterocolitis of Newborn; Risk Factors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NEC Group: All Premature Neonates born in Nancy and Lyon over 10 years and presenting with Necrotizing Enterocolitis
  Interventions: Other: Observation of related perinatal factors
- Control Group: All Premature Neonates born in Nancy and Lyon over 10 years without Necrotizing Enterocolitis throughout the neonatal period
  Interventions: Other: Observation of related perinatal factors

INTERVENTIONS:
Other: Observation of related perinatal factors — Data described in Primary outcome measures will be collected in both groups

SUMMARY:
With premature newborn increase survival, the risk of serious neonatal morbidity, such as necrotizing enterocolitis (NEC), also increased. NEC affects between 2 to 7% of premature infants including 5 to 22% of newborns weighing less than 1000 g.

NEC is an acquired disease, caused by inflammation of the intestinal lining. It is the most common life-threatening gastrointestinal emergency of prematurity, associated with a significant morbidity and mortality.

The etiology and physiopathology are multifactorial, complex, and remain poorly understood. The mechanism of the lesions seems to involve factors including immaturity of the intestinal barrier and the immune system, microvascular imbalance, disturbed gut flora and systemic inflammation.

Despite improved knowledge about this disease, the proportion of surviving patients has not improved for several years. It frequently leads to long-term sequelae depending on the severity of the NEC and its treatment.

Early diagnosis and early treatment of NEC may reduce the risk of mortality and morbidity. The aim of this retrospective bi-centric study is to look for risk factors allowing the prediction of NEC in order to prevent and improve the early management of this disease.

ELIGIBILITY:
Inclusion Criteria:

* Premature newborns (< 37 weeks of gestation) having done a necrotizing enterocolitis stage II or III according to Bell's criteria.

Exclusion Criteria:

* Children term born (> 37 weeks of gestation)
* Necrotizing enterocolitis during an hospitalisation outside the NICU of Nancy or Lyon
* Malformation or pre-existing digestive pathology
* Complex or severe malformative pathologies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Premature newborns (< 37 weeks of gestation) having done a necrotizing enterocolitis stage II or III according to Bell's criteria.
  * Premature newborns (< 37 weeks of gestation) having grown up without nectrotizing enterocolitis at the same period of time, in order to associate 2 witness patient to one case patient.
Sampling Method: Non-Probability Sample
Enrollment: 459 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Necrotizing enterocolitis (NEC) | 10 years
  Number of infants with NEC at a Bell stage > 1 in Nancy as compared to Lyon
Risk factor of NEC during Pregnancy | 10 years
  Number of infants who had abnormal pregnancy course in each group (defined as the presence of multiple pregnancy; gestational hypertension; Intrauterine Growth Retardation defined as a birth weight below the 10th Centile of Fenton Curves; Abnormal heart rate at the time of delivery)
Gestational age of infants with NEC | 10 years
  Gestational age in weeks of infants presenting with NEC in Nancy as compared to Lyon

SECONDARY OUTCOMES:
Perinatal risk factor of NEC | 10 years
  Number of infants who did not receive antenatal maturation by steroids in Nancy as compared to Lyon
Place of birth as risk factor for NEC | 10 years
  Number of outborn infants in Nancy as compared to Lyon
Asphyxia at birth | 10 years
  Number of infants with an APGAR score < 7 in Nancy as compared to Lyon
NEC occurrence | 10 years
  Age of NEC onset in Nancy as compared to Lyon
Gender | 10 years
  Rate of baby boys presenting NEC in Nancy as compared to Lyon
Patent Ductus Arteriosus (PDA) | 10 years
  Number of enfants presenting a PDA requiring treatment in Nancy as compared to Lyon
Feeding | 10 years
  Number of infants for each Type of milk at the point of date in Nancy as compared to Lyon (Mothers own milk versus milk bank versus formula )
Infection | 10 years
  Number of infants treated for infection in Nancy as compared to Lyon
Red Blood Cell transfusion | 10 years
  Number of infants who required a transfusion before the occurence of NEC in Nancy as compared to Lyon

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Maternite Regionale Universitaire CHRU NANCY, Nancy, Lorraine
  - CHU LYON, Bron